CLINICAL TRIAL: NCT00132223
Title: Effects on the Diagnostic Accuracy of Magnetic Imaging Angiographies of the Supra-Aortic Vessels by Three Different Magnetic Resonance Contrast Agents in Patients With Headache and Dizziness or Epilepsy and Clinical Indication for an Angiography by Magnetic Imaging
Brief Title: Effects on the Diagnostic Accuracy of Magnetic Imaging Angiographies of the Supra-Aortic Vessels by Three Different Magnetic Resonance Contrast Agents in Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0710/2004-IKR
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2006-04-12 (Estimated); Status verified 2006-04

CONDITIONS: Headache; Epilepsy; Dizziness
Keywords: magnetic imaging; angiography; contrast agent; signal/noise ratio; contrast/noise ratio; vessel
MeSH Terms: conditions — Headache; Epilepsy; Dizziness | interventions — Contrast Media

INTERVENTIONS:
Drug: Contrast agent

SUMMARY:
Angiographies of the supra-aortic vessels by magnetic imaging have become common recently. So it was the purpose of this study to evaluate the imaging potential of different contrast agents.

Three contrast agents for magnetic resonance imaging are compared in angiographies of the supra-aortic arteries in a intraindividual study of 10 patients.

All applications of these contrast agents are performed with a flow of 2 ml/s. One contrast medium is applicated a second time with a reduced flow of 1 ml/s.

The angiographies of the supra-aortic vessels are evaluated by two experienced readers in a consensus reading. The signal/noise- and contrast/noise-ratio of anatomic vessel segments of the carotic and vertebral arteries are measured and compared to each other.

ELIGIBILITY:
Inclusion Criteria:

* Headache
* Epilepsia
* Dizziness

Exclusion Criteria:

* Pregnancy
* Metal implants (e.g. pacemaker)
* Contraindication for contrast agent
* Multiple allergies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10
Dates: Start 2005-04; Study Completion 2005-12

PRIMARY OUTCOMES:
intensity of vessels, muscle, air

SECONDARY OUTCOMES:
signal/noise ratio
contrast/nose ratio

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Tombach, MD, Study Chair — University of Muenster, Dept. of Clinical Radiology
Locations (1):
- University of Muenster, Dept. of Clinical Radiology, Münster, Germany